CLINICAL TRIAL: NCT02666742
Title: SafeTy and Efficacy of Direct Oral Anticoagulant Versus Aspirin for Reduction Of RisK of CErebrovascular Events in Patients Undergoing Ventricular Tachycardia Ablation (STROKE-VT)
Brief Title: DOACs for Stroke Prevention Post Ventricular Tachycardia Ablation
Acronym: STROKE-VT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kansas City Heart Rhythm Institute (Other)
Collaborators: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003241; CV185-415 (Other: KCHRF)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2021-08

CONDITIONS: Ventricular Tachycardia; Premature Ventricular Contraction; Stroke
Keywords: Radiofrequency ablation; anticoagulation; Direct oral anticoagulants; Aspirin; Ventricular arrhythmia
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes; Stroke | interventions — Rivaroxaban; Dabigatran; edoxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DOAC (Direct Oral Anticoagulant) (Experimental): Participants will be asked to take standard dose approved for stroke prophylaxis
  Interventions: Drug: DOAC
- Aspirin (Active Comparator): Participants will be asked to take 81 milligrams by mouth once per day.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: DOAC — DOAC is a blood thinning drug, also called direct oral anticoagulant. These group of drugs are approved by the U.S. Food and Drug Administration (FDA) for the treatment of stroke prophylaxis in atrial fibrillation and deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
  Other Names: Direct Oral Anti Coagulants; Rivaroxaban; Apixiban; Dabigatran; Edoxaban
  Arms: DOAC (Direct Oral Anticoagulant)
Drug: Aspirin — Aspirin works by reducing substances in the body that cause pain, fever, and inflammation. Aspirin is used to treat pain, and reduce fever or inflammation.
  Arms: Aspirin

SUMMARY:
The purpose of this study is to learn if taking a drug called direct oral anticoagulant after an ablation procedure keeps blood clots from forming and lowers the chance of having a stroke in patients with ventricular tachycardia or arrhythmia (VT).

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) or fast heart rhythm is a condition where the lower chambers (ventricles) of the heart beat too fast. This condition can be life threatening because these ventricles are the main pumping chambers of the heart. The fast heartbeat is caused by electrical impulses that travel incorrectly in your heart.

One way to treat VT is to have a catheter ablation procedure. A catheter ablation is a procedure that creates scar tissue in the heart to interrupt the electrical impulses that create irregular heart rhythms.

It is possible that the ablation procedure might cause a blood clot to form. The blood clot can stop blood flow to the brain and cause a stroke. When blood flow is interrupted to a certain part of the brain, that part does not receive enough oxygen. As a result of the stroke the affected areas of the brain are unable to function normally.

Direct oral anticoagulant (DOAC) is a blood thinning drug, also called an anticoagulant. It interferes with the body's natural blood clotting ability by inactivating a specific enzyme that the body needs to form blood clots.

Participation in this study will last about 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiofrequency catheter ablation for scar VT which includes VT secondary to ischemic cardiomyopathy and non-ischemic cardiomyopathy
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with Apixaban plus 33 days post-treatment completion
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and for a total of 93 days post-treatment completion
* Participants must agree to the use of one approved method of contraception

Exclusion Criteria:

* History of cerebral vascular accident/transient ischemic attack (CVA/TIA) in last 3 months
* Cardiac surgery or neurosurgery within 3 months of the intended procedure date
* Any active bleeding
* Severe hypersensitivity reaction to ELIQUIS (including drug hypersensitivity, such as skin rash and allergic reactions)
* Participants cannot have prosthetic heart valves
* History or bleeding and clotting disorders
* Contraindications to Aspirin therapy
* Contraindication to oral anticoagulation
* Patient on an anticoagulant prior to the ablation for other primary indications like atrial fibrillation (AF), deep vein thrombosis (DVT) or a mechanical valve
* Evidence of intracardiac thrombus
* Patient with Creatinine Clearance of < 30 cc/min
* Participation in another investigational study related to oral anticoagulation, drug and/or device intervention
* Claustrophobic patients
* Implantable Cardioverter Defibrillator (ICD) generator placement before the year 2000
* Has an ICD and is pacing dependent without underlying rhythm upon interrogation at baseline
* Patient has abandoned leads
* Patients who are on p-glycoprotein inducers or inhibitors where the dose of Apixaban cannot be effectively altered

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Research Foundation
Locations (5):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - KCHRF, Overland Park, Kansas
  - Montefiore Medical Center, The Bronx, New York
  - TCAI, Austin, Texas
- Jayadeva Institute of Medical Sciences, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabral KP, Ansell JE. The role of factor Xa inhibitors in venous thromboembolism treatment. Vasc Health Risk Manag. 2015 Jan 30;11:117-23. doi: 10.2147/VHRM.S39726. eCollection 2015. PMID 25673997
- [Background] Ghanbari H, Baser K, Jongnarangsin K, Chugh A, Nallamothu BK, Gillespie BW, Baser HD, Suwanagool A, Crawford T, Latchamsetty R, Good E, Pelosi F Jr, Bogun F, Morady F, Oral H. Mortality and cerebrovascular events after radiofrequency catheter ablation of atrial fibrillation. Heart Rhythm. 2014 Sep;11(9):1503-11. doi: 10.1016/j.hrthm.2014.05.003. Epub 2014 May 6. PMID 24813379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women (with negative urine pregnancy test or non-breastfeeding) aged at least 18 years old were eligible for the study if they underwent radiofrequency ablation (RFA) for VT (secondary to ischemic or nonischemic cardiomyopathy) or PVC's.
Groups:
- Direct Oral Anticoagulant (DOAC): Participants will be asked to take a DOAC (Rivaroxaban/Apixiban/Dabigatran/Edoxaban) dose that is approved for stroke prophylaxis for 30 days post ablation
  DOAC: DOAC is a blood thinning drug, also called an anticoagulant. DOAC is approved by the U.S. Food and Drug Administration (FDA) for the prophylaxis of stroke in atrial fibrillation patients and treatment of deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
Period: Overall Study
Arm/Group | Direct Oral Anticoagulant (DOAC) | Aspirin
Started | 123 | 123
Completed | 123 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing VT or PVC ablation are enrolled into the study. Baseline characteristics of patients including demographics, comorbidities, cardiac function etc were collected and analyzed
Groups:
- DOAC: Participants will be asked to take approved dose of the drug for stroke Px
  DOAC Apixaban is a blood thinning drug, also called an anticoagulant. DOAC is approved by the U.S. Food and Drug Administration (FDA) for stroke prophylaxis and the treatment of deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
- Total: Total of all reporting groups
Arm/Group | DOAC | Aspirin | Total
Number analyzed (Participants) | 123 | 123 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (12.5) | 58.3 (14.7) | 59.95 (13.7438)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 99 | 104 | 203
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Anti-arrhythmic drugs [Count of Participants; unit: Participants] | 100 | 90 | 190

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Transient Ischemic Attack
Description: Transient ischemic attack(TIA) - defined as a transient episode of neurological dysfunction caused by focal brain, spinal cord, or retinal ischemia, without acute infarction.
Time Frame: First 30 days of post ablation
Population: this is a population group undergoing VT or premature ventricular contraction (PVC) ablation
Measure: Number; unit: participants
Groups:
- DOAC: DOAC is a blood thinner group
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
participants | 6 | 22
Statistical Analysis 1: Comparison: DOAC vs Aspirin; Due to lack of precedent robust clinical data, we performed exploratory study to evaluate safety and efficacy of DOAC vs. Aspirin (ASA) in patients undergoing left ventricular arrhythmia (LVA) ablation; therefore, sample size calculation was not undertaken; Test type: Superiority — Continuous variables were compared by two-sample t-tests and categorical variables by chi-square test. All tests were two-tailed, and a P value less than 0.05 was considered to indicate statistical significance. Bonferroni correction was not performed due to prespecified outcomes in the trial. Analyses were performed using GraphPad 6; p = 0.001, Chi-squared

2. Primary Outcome: Number of Participants With Stroke
Description: Stroke - incidence of ischemic stroke - defined as an episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction.
Time Frame: First 30 days of post ablation
Population: This is a population group undergoing VT or PVC ablation
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 0 | 8

3. Primary Outcome: Number of Participants With Asymptomatic Cerebral Event on MRI - 24 Hours
Description: MRI detected asymptomatic cerebrovascular events (ACE) at 24 hours.
Time Frame: 24 Hours post ablation
Population: This is a population group undergoing VT or PVC ablation
Measure: Count of Participants; unit: Participants
Groups:
- DOAC: Participants will be asked to take standard dose approved for stroke prophylaxis
  DOAC: DOAC is a blood thinning drug, also called direct oral anticoagulant. These group of drugs are approved by the U.S. Food and Drug Administration (FDA) for the treatment of stroke prophylaxis in atrial fibrillation and deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 15 | 28

4. Primary Outcome: Number of Participants With Asymptomatic Cerebral Event on MRI - 30 Days
Description: MRI detected asymptomatic cerebrovascular events (ACE) at 30 days follow-up.
Time Frame: 24 Hours to 30 days of post ablation
Population: This is a population group undergoing VT or PVC ablation
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 8 | 22

5. Secondary Outcome: Number of Participants With Acute Procedure Related Complications
Description: The secondary endpoints included procedure-related complications (composite of any vascular complication, pericardial complication, heart block, thromboembolic event excluding stroke or TIA) and in-hospital mortality.
Time Frame: Day 30
Population: patients who meet inclusion criteria
Measure: Count of Participants; unit: Participants
Groups:
- DOAC: Participants will be asked to take DOAC as prescribed
  DOAC is a blood thinning drug, also called an anticoagulant. DOACs are approved by the U.S. Food and Drug Administration (FDA) for stroke prophylaxis and the treatment of deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 15 | 17

6. Secondary Outcome: Number of Participants With Cardiac Tamponade
Description: Cardiac tamponade is a medical emergency that takes place when abnormal amounts of fluid accumulate in the pericardial sac compressing the heart and leading to a decrease in cardiac output and shock.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 4 | 3

7. Secondary Outcome: Number of Participants With Fatal Pulmonary Embolism
Description: A pulmonary embolism is a blood clot in the lung that occurs when a clot in another part of the body (often the leg or arm) moves through the bloodstream and becomes lodged in the blood vessels of the lung. This restricts blood flow to the lungs, lowers oxygen levels in the lungs and increases blood pressure in the pulmonary arteries.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 0 | 1

8. Secondary Outcome: Number of Participants With Progressive Heart Failure and Electromechanical Dissociation (EMD)
Description: Heart failure means that the heart isn't pumping as well as it should be.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 4 | 4

9. Secondary Outcome: Number of Participants With Groin Hematoma
Description: A hematoma is a collection of blood outside of a blood vessel.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 3 | 4

10. Secondary Outcome: Number of Participants With Retroperitoneal Bleed
Description: Retroperitoneal bleeding occurs when blood enters into space immediately behind the posterior reflection of the abdominal peritoneum. The organs of this space include the esophagus, aorta, inferior vena cava, kidneys, ureters, adrenals, rectum, parts of the duodenum, parts of the pancreas, and parts of the colon.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 2 | 2

11. Secondary Outcome: Number of Participants With Heart Block
Description: Heart block is a type of heart rhythm disorder (arrhythmia). It is the slowing down or interruption of the electrical signal from the upper chambers of the heart (the atria) to the lower chambers (the ventricles). The electrical signal causes the heart muscle to contract and the heart to beat.
Time Frame: Day 30
Population: Patients who meet inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 2 | 3

12. Secondary Outcome: Number of Participants With In-hospital Mortality
Description: Death occurring during the hospital stay.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | DOAC | Aspirin
Number analyzed (Participants) | 123 | 123
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: First 30 days of post ablation
Groups:
- Apixaban: Participants will be asked to take 5 milligrams by mouth twice per day.
  Apixaban: Apixaban is a blood thinning drug, also called an anticoagulant. Apixaban is approved by the U.S. Food and Drug Administration (FDA) for the treatment of deep vein thrombosis and pulmonary embolism, which are blood clots in the veins or lungs.
Arm/Group | Apixaban | Aspirin
All-Cause Mortality (participants affected / at risk) | 5/123 | 3/123
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/123
Other Adverse Events (participants affected / at risk) | 0/123 | 0/123

LIMITATIONS AND CAVEATS:
Our results should be considered in light of several significant limitations. An important limitation was the lack of long-term follow-up and quality-of-life and neurocognitive function information. Another methodological limitation of the outcomes was that the ASA group did not get a loading dose, perhaps the delay in achieving the therapeutic effects in denovo ASA initiation could increase the risk of events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02666742/Prot_SAP_000.pdf